CLINICAL TRIAL: NCT06313840
Title: Central Sleep Apnea Prevalence and Impact on Cognitive Function in Patients With Heart Failure With Reduced or Mildly Reduced Left Ventricular Ejection Fraction
Acronym: COG01
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP3125
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Central Sleep Apnea
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Case group - subjects with central sleep apnea: Patients with moderate to severe CSA defined by an apnea hypopnea index (AHI) ≥ 15 events per hour and a central apnea hypopnea index (CAHI) ≥ 50% of total AHI.
- Control group - subjects with no sleep disordered breathing: Patients with no SDB defined by an AHI < 5 events per hour.
- Other SDB group - subjects with other forms of sleep disordered breathing: Patients that do not meet criteria for CSA or no SDB

SUMMARY:
Study to assess the prevalence of central sleep apnea in patients with heart failure with reduced or mildly reduced left ventricular ejection fraction (LVEF <50%) followed by case-control study to assess the link between central sleep apnea and cognitive function

DETAILED DESCRIPTION:
The study will be conducted in two phases: prevalence phase and cognitive phase.

Adult patients with HFrEF/HFmrEF will perform a home sleep apnea test (HSAT). Patients will be assigned to one of the following groups based on their sleep study results: CSA, other SDB, or no SDB. This constitutes the prevalence phase of the study.

The cognitive phase of the study is a case-control study that will assess cognitive function in 20 patients in the CSA group (case) and 20 patients in the no SDB group (control).

ELIGIBILITY:
Prevalence Phase Inclusion Criteria:

1. Diagnosed with heart failure with reduced or mildly reduced left ventricular ejection fraction (LVEF <50%) at least 3 months prior to enrollment
2. New York Heart Association (NYHA) functional class II-IV
3. Treated and optimized on heart failure guideline directed medical therapy as indicated for at least 4 weeks, including angiotensin receptor-neprilysin inhibitors (ARNI) (or angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blocker (ARB)), aldosterone receptor antagonists, beta-blockers and/or sodium glucose co-transporter 2 (SGLT-2) antagonists
4. Age 50 years or older
5. Signed Institutional Review Board (IRB) or Ethics Committee (EC) approved informed consent
6. In the opinion of the investigator, subject is willing and able to comply with the protocol, including the cognitive function assessment

Prevalence Phase Exclusion Criteria:

1. Hospitalized for heart failure-related complications in the last 4 weeks
2. History of SDB and/or prior or ongoing treatment for SDB or tested for SDB within the prior year

Cognitive Phase Inclusion Criteria:

1. AHI ≥ 15 events per hour and CAHI ≥ 50% of total AHI (Case group) or AHI < 5 events per hour (Control group) based on the baseline HSAT
2. Per the patient and investigator, willing and able to postpone CSA treatment until completion of the study assessment visit (Visit 3)

Cognitive Phase Exclusion Criteria:

1. Color blindness
2. Currently taking opioids
3. Has taken medications for memory/cognition within the last 3 months (including but not limited to cholinesterase inhibitors and/or glutamate regulators)
4. Cerebrovascular accident (stroke or transient ischemic attack) in the last 12 months
5. Diagnosed with neurological disease including but not limited to history of seizures, meningitis, traumatic brain injury, amyotrophic lateral sclerosis, multiple sclerosis, attention-deficit/hyperactivity disorder (ADHD) or autism.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 50 years or older with HFrEF/HFmrEF and no history of sleep disordered breathing (SDB) and not tested for SDB within the prior year will be tested for sleep apnea using a home sleep apnea test (WatchPAT device).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of CSA in tested HFrEF/HFmrEF patients | Through study completion, an average of 1 year
  Determine the prevalence of CSA in a contemporary population of HFrEF/HFmrEF patients completing a Home Sleep Apnea Test (using a WatchPAT device) during the prevalence phase of the study.

SECONDARY OUTCOMES:
Difference in cognitive function scores between the HFrEF/HFmrEF CSA and no SDB groups using the CANTAB assessment. | Through study completion, an average of 1 year
  Evaluate differences in cognitive function between adult patients with heart failure with reduced or mildly reduced left ventricular ejection fraction (HFrEF/HFmrEF) (LVEF <50%) and central sleep apnea (CSA) versus patients with HFrEF/HFmrEF and no sleep disordered breathing (SDB) using a battery of assessments from the Cambridge Neuropsychological Test Automated Battery (CANTAB).

CONTACTS AND LOCATIONS:
Overall Officials: Kathy McPherson, Study Director — ZOLL Respciardia
Locations (1):
- Szpital Uniwersytecki we Wrocławiu, Wroclaw, Poland